CLINICAL TRIAL: NCT00900341
Title: LABORATORY STUDIES OF SOFT TISSUE SARCOMAS
Brief Title: Studying Tumor Tissue Samples From Patients With Soft Tissue Sarcoma
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 05-0509-04; P30CA023074 (NIH); UARIZ-HSCA0535 (Other: CDR0000597591); UARIZ-17879
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Sarcoma
Keywords: adult soft tissue sarcoma; childhood soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor tissue samples from patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a pilot program for the collection, archiving, and experimental analyses of soft tissue sarcomas (STS).
* To obtain STS tumors from cancer patients undergoing tumor removal or core needle biopsies.
* To evaluate cellular and molecular factors involved in STS oncogenesis by studying samples derived from human tumor specimens.
* To develop an accompanying bioinformatics database of the demographics of STS patients from which tumor specimens are derived for experimental study.

OUTLINE: Tumor tissue samples are analyzed for gene and protein expression by cDNA microarray analysis, RT-PCR, immunohistochemistry, in vitro transformation assays, RNA interference, and Western blot or immunoprecipitation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Patients with soft tissue sarcoma (STS) undergoing evaluation, treatment, and/or follow-up at the Arizona Cancer Center or University Medical Center
  * Patients undergoing surgical treatment for STS removal or core needle biopsy for medically indicated diagnostic or therapeutic purposes

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical treatment for soft tissue sarcomas removal or core needle biopsy for medically indicated diagnostic or therapeutic purposes.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identification of molecular targets that would improve the diagnosis, prognosis, and/or treatment of STS | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee D. Cranmer, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States